CLINICAL TRIAL: NCT04425850
Title: USEFULNESS of Topic Ivermectin and Carrageenan to Prevent Contagion of Covid Among Healthy People and Health Personnel
Brief Title: USEFULNESS of Topic Ivermectin and Carrageenan to Prevent Contagion of Covid 19
Acronym: IVERCAR
Status: Completed | Type: Observational
Sponsor: Eurnekian Public Hospital (Other)
Responsible Party: Principal Investigator, Hector E Carvallo, Principal Investigator, Eurnekian Public Hospital
Other Study IDs: IVERCAR
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: IVERMECTIN CARRAGEENAN COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IVER+: Adults, both genders, no age limit. They will be provided with topical medication, to be used 5 times a day. They will follow standard prophylactic measures and use PPE as suggested by OMS.
  Interventions: Combination Product: Iota carrageenan nasal spray and Ivermectin oral drops (used as buccal drops)
- IVER-: Adults, both genders, no age limit They will follow standard prophylactic measures and use PPE suggestions, only.

INTERVENTIONS:
Combination Product: Iota carrageenan nasal spray and Ivermectin oral drops (used as buccal drops) — Topical application in the nose and oral cavity
  Other Names: Nasitral (iota carrageenan nasal spray), Ivercass (ivermectin oral drops)
  Groups: IVER+

SUMMARY:
Estimation of the prevalence and contagiousness of undocumented novel coronavirus infections is critical for understanding the overall prevalence and pandemic potential of this disease.

It is estimated that 86% of all infections were undocumented [95% credible interval (CI): 82-90%] before the 23 January 2020 travel restrictions. The transmission rate of undocumented infections per person was 55% the transmission rate of documented infections (95% CI: 46-62%), yet, because of their greater numbers, undocumented infections were the source of 79% of the documented cases.

Ivermectin + Carrageenan, taking advantage of their virucidal effects, are aimed at reducing the contagion.

DETAILED DESCRIPTION:
CONTAGION COURSE Estimation of the prevalence and contagiousness of undocumented novel coronavirus infections is critical for understanding the overall prevalence and pandemic potential of this disease.

Observations of reported infection within China, in conjunction with mobility data, a networked dynamic metapopulation model, and Bayesian inference, to infer critical epidemiological characteristics associated with SARS-CoV-2, including the fraction of undocumented infections and their contagiousness, have been attempted. The rapid geographic spread of SARS-CoV-2 indicate that containment of this virus will be particularly challenging.

DISSEMINATION BY DROPLETS For COVID-19, the salivary gland could be an important source of the virus in saliva and would generate infectious saliva on a sustained basis.

ACE2 expression in the minor salivary glands was higher than in the lungs, suggesting that the salivary glands is a potential target for COVID-19.

The positive rate of COVID-19 in the patients' saliva can reach 91.7%, and the saliva samples can also culture the live virus.

In addition to mobility restrictions of people, the World Health Organization and the Governments have prescribed maintaining an inter-personal distance of 1.5 or 2 m (about 6 feet) from each other in order to minimize the risk of contagion through the droplets that we usually disseminate around us from nose and mouth. However, recently published studies support the hypothesis of virus transmission over a distance of 2 m from an infected person. Researchers have proved the higher aerosol and surface stability of SARS-COV-2 as compared with SARS-COV-1 (with the virus remaining viable and infectious in aerosol for hours) and that airborne transmission of SARS-CoV can occur besides close-distance contacts. Indeed, there is reasonable evidence about the possibility of SARS-COV-2 airborne transmission due to its persistence into aerosol droplets in a viable and infectious form. Based on the available knowledge and epidemiological observations, it is plausible that small particles containing the virus may diffuse in indoor environments covering distances up to 10 m from the emission sources, thus representing a kind of aerosol transmission. On-field studies carried out inside Wuhan Hospitals showed the presence of SARS-COV-2 RNA in air samples collected in the hospitals and also in the surroundings, leading to the conclusion that the airborne route has to be considered an important pathway for viral diffusion. Similar findings are reported in analyses concerning air samples collected at the Nebraska University Hospital. On March 16th, we have released a Position Paper emphasizing the airborne route as a possible additional factor for interpreting the anomalous COVID-19 outbreaks in northern Italy, ranked as one of the most polluted areas in Europe and characterized by high particulate matter (PM) concentrations. The available information on the SARS-COV-2 spreading supports the hypothesis of airborne diffusion of infected droplets from person to person at a distance greater than two meters (6 feet). The inter-personal distance of 2 m can be reasonably considered as an effective protection only if everybody wears face masks in daily life activities.

IVERMECTIN CONCENTRATION IN SALIVARY GLANDS The concentration of ivermectin was tested in different tissues, in different studies, both in animals and human beings. The concentration in salivary glands proved to be adequately acceptable.

CARRAGEENAN VIRUCIDAL EFFECTS Iota Carrageenan is widely used in gastronomic, cosmetic and pharmacologic industry.

Recently, its intrinsic virucidal effectas were proved over a variety of virus (herpes simplex, Japanese Encephalitis, Rhinovirus, etc.).

Its mechanism of action is preventing virus adsorption to host cells. By applying both drugs topically, 5 times per day, in nasal and oral mucosae, we try to reduce contagion.

ELIGIBILITY:
Inclusion criteria

1. Not younger than 18 years of either sex
2. Health personnel from the Dr. Alberto Eurnekian Interzonal University Hospital
3. No COVID-19 related symptoms
4. Able to understand and give written informed consent

Exclusion criteria

1. Known hypersensitivity or allergy to any component of the product under evaluation
2. Age under 18 years
3. Use of immunosuppressants (including systemic corticosteroids) in the past 30 days.
4. Pregnant or nursing.
5. Patients with other acute infectious diseases.
6. Patients with autoimmune disease and / or decompensated chronic diseases.
7. Unable to fulfill the administrative tasks proposed by the study.
8. Infection with SARSCoV-2 confirmed by PCR or rapid test authorized by ANMAT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers testing negative for COVID-19 just before inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Eurnekian, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Harden EA, Falshaw R, Carnachan SM, Kern ER, Prichard MN. Virucidal activity of polysaccharide extracts from four algal species against herpes simplex virus. Antiviral Res. 2009 Sep;83(3):282-9. doi: 10.1016/j.antiviral.2009.06.007. Epub 2009 Jul 1. PMID 19576248
- [Background] Carlucci MJ, Scolaro LA, Noseda MD, Cerezo AS, Damonte EB. Protective effect of a natural carrageenan on genital herpes simplex virus infection in mice. Antiviral Res. 2004 Nov;64(2):137-41. doi: 10.1016/j.antiviral.2004.07.001. PMID 15498610
- [Background] Ashraf S, Prichard R. Ivermectin exhibits potent anti-mitotic activity. Vet Parasitol. 2016 Aug 15;226:1-4. doi: 10.1016/j.vetpar.2016.06.015. Epub 2016 Jun 11. PMID 27514873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Health personnel
Pre-assignment Details: Once consent was signed, compliance with all the eligibility criteria verified, and inclusion of the subject decided, the investigator assigns corresponding treatment according to the randomization carried out.
  It includes volunteers for both cohorts, provided they have test negative for COVID 19 in swabs obtained immediately before inclusion.
Groups:
- IVER+: Standard prophylactic measures and PPEs + iota carrageenan (nasal and buccal) and ivermectin (buccal)
- IVER-: Standard prophylactic measures and PPE only
Period: Overall Study
Arm/Group | IVER+ | IVER-
Started | 131 (Standard prophylactic measures and PPE + iota carrageenan (nasal and buccal) and ivermectin (buccal)) | 98 (Standard prophylactic measures and PPE only)
Completed | 131 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IVER+: Adults, both genders, no age limit. They will be provided with topical medication, to be used 5 times a day. PPEs used as suggested by OMS.
  iota carrageenan: topical use on nasal mucosae
  Ivermectin: Topical use on oral mucosae
- IVER-: Same as IVER+ They will follow PPEs suggestions, only.
- Total: Total of all reporting groups
Arm/Group | IVER+ | IVER- | Total
Number analyzed (Participants) | 131 | 98 | 229
Age, Continuous [Median (Full Range); unit: years] | 42 [25 to 60] | 39 [28 to 50] | 40 [25 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 72 | 142
  Male | 61 | 26 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 131 | 98 | 229
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 131 | 98 | 229
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 131 | 98 | 229

OUTCOME MEASURES:

1. Primary Outcome: Number of Infected Subjects
Description: Number of participants testing positive for COVID-19 after inclusion in each arm
Time Frame: 28 days
Population: Hispanic
Measure: Count of Participants; unit: Participants
Groups:
- IVER+: Standard prophylactic measures and PPEs + topical treatment with iota carrageenan (nasal and buccal) and ivermectin (buccal)
- IVER-: Standard prophylactic measures and PPEs only
Arm/Group | IVER+ | IVER-
Number analyzed (Participants) | 131 | 98
Participants | 0 | 11
Statistical Analysis 1: Comparison: IVER+ vs IVER-; Chi-squared test on the percentage of subjects who contracted COVID-19 in each arm; Test type: Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Adverse Events Other Than Those Resulting From Contagion or Disease Progression
Description: Adverse events reported by subjects of each arm are recorded other than those resulting from contagion or disease progression
Time Frame: 28 days
Population: Hispanic
Measure: Count of Participants; unit: Participants
Groups:
- IVER+: Standard prophylactic measures and PPE + Treatment with iota carragenan (nasal and buccal) and ivermectin (buccal only)
Arm/Group | IVER+ | IVER-
Number analyzed (Participants) | 131 | 98
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Medical examination Chart of adverse events filled in by subjects
Arm/Group | IVER+ | IVER-
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/98
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/98
Other Adverse Events (participants affected / at risk) | 0/131 | 11/98
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVER+ (N=131) | IVER- (N=98)
Contagion (Infections and infestations) | 0 (0) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT04425850/Prot_SAP_000.pdf